CLINICAL TRIAL: NCT00906698
Title: Phase I Open Label Trial to Assess Safety of BIBW 2992 With Vinorelbine in Solid Tumors Known to Overexpress HER2 and/or EGFR
Brief Title: Afatinib and Vinorelbine in Tumours Known to Overexpress EGFR and/or HER2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1200.69; 2008-006290-32 (EudraCT Number: EudraCT)
Record Dates: First submitted 2009-05-14; First posted 2009-05-21 (Estimated); Results first posted 2014-04-17 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-03

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

ARMS (2):
- BIBW 2992 and vinorelbine i.v (Experimental): Daily low (20mg), medium (40mg) and high (50mg) dosages of BIBW 2992 with standard dosage of vinorelbine i.v.
  Interventions: Drug: BIBW 2992 low (20mg) dosage; Drug: BIBW 2992 medium (40mg) dosage; Drug: BIBW 2992 high (50mg) dosage; Drug: Vinorelbine i.v. 25 mg/m²
- BIBW 2992 and vinorelbine per os (Experimental): Daily low (20mg), medium (40mg) and high (50mg) dosages of BIBW 2992 with standard dosage of vinorelbine per os.
  Interventions: Drug: BIBW 2992 low (20mg) dosage; Drug: BIBW 2992 medium (40mg) dosage; Drug: BIBW 2992 high (50mg) dosage; Drug: Vinorelbine per os 60 mg/m²; Drug: Vinorelbine per os 80 mg/m²

INTERVENTIONS:
Drug: BIBW 2992 low (20mg) dosage — Patients will receive 20mg dosage per day of BIBW 2992 plus standard dosage of vinorelbine.
Drug: BIBW 2992 medium (40mg) dosage — Patients will receive 40mg dosage per day of BIBW 2992 plus standard dosage of vinorelbine.
Drug: BIBW 2992 high (50mg) dosage — Patients will receive 50mg dosage of BIBW 2992 plus standard dosage of vinorelbine.
Drug: Vinorelbine per os 60 mg/m² — Patients will receive 60 mg/m² Vinorelbine per os at J1 J8 and J15
  Arms: BIBW 2992 and vinorelbine per os
Drug: Vinorelbine per os 80 mg/m² — Patients will receive 80 mg/m² Vinorelbine per os at J22
  Arms: BIBW 2992 and vinorelbine per os
Drug: Vinorelbine i.v. 25 mg/m² — Patients will receive 25 mg/m² of Vinorelbine i.v.
  Arms: BIBW 2992 and vinorelbine i.v

SUMMARY:
To determine the maximum tolerated dose, safety, pharmacokinetics and anti-tumour efficacy of oral BIBW 2992 in combination with intravenous or oral vinorelbine

ELIGIBILITY:
Inclusion criteria:

* Histologically or cytologically confirmed diagnosis of malignancy that is now advanced, non resectable and/or metastatic
* Tumours historically known to overexpress EGFR and/or HER2

Exclusion criteria:

* Prior treatment with HER2 inhibiting drugs within the past 4 weeks before the start of therapy or concomitantly with this trial.
* Prior treatment with EGFR inhibiting drugs within the past two weeks before the start of therapy or concomitantly with this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2009-06; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (2):
- France (2):
  - 1200.69.3301 Boehringer Ingelheim Investigational Site, Toulouse
  - 1200.69.3302 Boehringer Ingelheim Investigational Site, Villejuif

RESULTS

PARTICIPANT FLOW:
Groups:
- Afatinib 20mg With Vinorelbine i.v.: Continuous daily dosing of Afatinib 20mg orally and weekly Vinorelbine 25 mg/m2 intravenously (days 1, 8, 15 and 22) in a 4-weekly course. Patients will be eligible for repeated treatment courses in the absence of clinical disease progression or undue toxicity
- Afatinib 40mg With Vinorelbine i.v.: Continuous daily dosing of Afatinib 40mg orally and weekly Vinorelbine 25 mg/m2 intravenously (days 1, 8, 15 and 22) in a 4-weekly course. Patients will be eligible for repeated treatment courses in the absence of clinical disease progression or undue toxicity.
- Afatinib 50mg With Vinorelbine i.v.: Continuous daily dosing of Afatinib 50mg orally and weekly Vinorelbine 25 mg/m2 intravenously (days 1, 8, 15 and 22) in a 4-weekly course. Patients will be eligible for repeated treatment courses in the absence of clinical disease progression or undue toxicity.
- Afatinib 20mg With Vinorelbine Per os: Continuous daily dosing of Afatinib 20mg orally and oral vinorelbine 60 mg/m2/week for days 1,8,15 of first cycle, and 80mg/m2 from day 22 first cycle onwards, weekly. Patients will be eligible for repeated treatment courses in the absence of clinical disease progression or undue toxicity .
- Afatinib 40mg With Vinorelbine Per os: Continuous daily dosing of Afatinib 40mg orally and oral vinorelbine 60 mg/m2/week for days 1,8,15 of first cycle, and 80mg/m2 from day 22 first cycle onwards, weekly. Patients will be eligible for repeated treatment courses in the absence of clinical disease progression or undue toxicity.
- Afatinib 50mg With Vinorelbine Per os: Continuous daily dosing of Afatinib 50mg orally and oral vinorelbine 60 mg/m2/week for days 1,8,15 of first cycle, and 80mg/m2 from day 22 first cycle onwards, weekly. Patients will be eligible for repeated treatment courses in the absence of clinical disease progression or undue toxicity.
Period: Overall Study
Arm/Group | Afatinib 20mg With Vinorelbine i.v. | Afatinib 40mg With Vinorelbine i.v. | Afatinib 50mg With Vinorelbine i.v. | Afatinib 20mg With Vinorelbine Per os | Afatinib 40mg With Vinorelbine Per os | Afatinib 50mg With Vinorelbine Per os
Started | 3 | 19 | 6 | 4 | 18 | 5
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 19 | 6 | 4 | 18 | 5
Not completed — Dose-limiting toxicity (DLT) | 0 | 6 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 2 | 0 | 4 | 1
Not completed — Disease progression | 3 | 12 | 4 | 4 | 12 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0
Not completed — incl. non compliance, lost to follow-up | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Afatinib 20mg With Vinorelbine Per os: Continuous daily dosing of Afatinib 20mg orally and oral vinorelbine 60 mg/m2/week for days 1,8,15 of first cycle, and 80mg/m2 from day 22 first cycle onwards, weekly. Patients will be eligible for repeated treatment courses in the absence of clinical disease progression or undue toxicity.
- Total: Total of all reporting groups
Arm/Group | Afatinib 20mg With Vinorelbine i.v. | Afatinib 40mg With Vinorelbine i.v. | Afatinib 50mg With Vinorelbine i.v. | Afatinib 20mg With Vinorelbine Per os | Afatinib 40mg With Vinorelbine Per os | Afatinib 50mg With Vinorelbine Per os | Total
Number analyzed (Participants) | 3 | 19 | 6 | 4 | 18 | 5 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (15.3) | 55.3 (8.0) | 61.7 (5.0) | 55.3 (6.2) | 50.9 (9.5) | 51.0 (8.3) | 54.4 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 11 | 4 | 0 | 11 | 4 | 31
  Male | 2 | 8 | 2 | 4 | 7 | 1 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLT)
Description: Number of participants with DLT for the determination of the Maximum Tolerated Dose (MTD). 3+3 dose escalation design. MTD based on DLTs during first treatment course. After MTD was determined, additional patients were included at the MTD in an expansion cohort.
Time Frame: 28 days
Population: Treated Set (TS). TS consisted of all patients who were dispensed study medication and have taken at least 1 dose of Afatinib.
Measure: Number; unit: participants
Arm/Group | Afatinib 20mg With Vinorelbine i.v. | Afatinib 40mg With Vinorelbine i.v. | Afatinib 50mg With Vinorelbine i.v. | Afatinib 20mg With Vinorelbine Per os | Afatinib 40mg With Vinorelbine Per os | Afatinib 50mg With Vinorelbine Per os
Number analyzed (Participants) | 3 | 19 | 6 | 4 | 18 | 5
participants
  First cycle (N=3;6;6;4;6;5) | 0 | 1 | 4 | 0 | 1 | 3
  Expansion cohort (N=0;13;0;0;12;0) | NA — no expansion cohort for this arm | 7 | NA — no expansion cohort for this arm | NA — no expansion cohort for this arm | 2 | NA — no expansion cohort for this arm

2. Secondary Outcome: Number of Patients With Best Overall Response
Description: Overall response is defined as complete response, partial response and stable disease and was assessed according to Response Evaluation Criteria in Solid Tumours (RECIST 1.0). Complete response (CR) and partial response (PR) had to be confirmed by a subsequent tumour assessment at least 28 days after the criteria for CR or PR were first met. To confirm a status of stable disease, the duration of stable disease was to be at least 42 days.
Time Frame: From first dose of study medication to response measurement, up to 44 months. Tumour assessments were performed at screening, week 8, week 16, week 24, and every 8 weeks thereafter.
Population: All patients from the Treated Set (TS).
Measure: Number; unit: participants
Arm/Group | Afatinib 20mg With Vinorelbine i.v. | Afatinib 40mg With Vinorelbine i.v. | Afatinib 50mg With Vinorelbine i.v. | Afatinib 20mg With Vinorelbine Per os | Afatinib 40mg With Vinorelbine Per os | Afatinib 50mg With Vinorelbine Per os
Number analyzed (Participants) | 3 | 19 | 6 | 4 | 18 | 5
participants
  Complete response | 0 | 0 | 0 | 0 | 0 | 0
  Partial response | 0 | 0 | 0 | 0 | 3 | 0
  Stable disease | 1 | 10 | 5 | 0 | 6 | 5
  Progressive disease | 2 | 6 | 0 | 4 | 7 | 0
  Missing | 0 | 3 | 1 | 0 | 2 | 0

3. Secondary Outcome: Number of Patients With Objective Response (OR)
Description: OR is defined as confirmed complete response and confirmed partial response (PR) and was assessed according to Response Evaluation Criteria in Solid Tumours (RECIST 1.0).
Time Frame: as for outcome 2
Population: All patients from the Treated Set (TS).
Measure: Number; unit: participants
Arm/Group | Afatinib 20mg With Vinorelbine i.v. | Afatinib 40mg With Vinorelbine i.v. | Afatinib 50mg With Vinorelbine i.v. | Afatinib 20mg With Vinorelbine Per os | Afatinib 40mg With Vinorelbine Per os | Afatinib 50mg With Vinorelbine Per os
Number analyzed (Participants) | 3 | 19 | 6 | 4 | 18 | 5
participants | 0 | 0 | 0 | 0 | 3 | 0

4. Secondary Outcome: Number of Patients With Disease Control (DC)
Description: DC is defined as confirmed complete response (CR), partial response (PR) and stable disease (SD) and was assessed according to Response Evaluation Criteria in Solid Tumours (RECIST 1.0).
Time Frame: as for outcome 2
Population: All patients from the Treated Set (TS).
Measure: Number; unit: participants
Arm/Group | Afatinib 20mg With Vinorelbine i.v. | Afatinib 40mg With Vinorelbine i.v. | Afatinib 50mg With Vinorelbine i.v. | Afatinib 20mg With Vinorelbine Per os | Afatinib 40mg With Vinorelbine Per os | Afatinib 50mg With Vinorelbine Per os
Number analyzed (Participants) | 3 | 19 | 6 | 4 | 18 | 5
participants | 1 | 10 | 5 | 0 | 9 | 5

5. Secondary Outcome: Time to Objective Response
Description: The time to OR was the duration from the first treatment to the time when the measurement criteria for first documented confirmed CR and/or PR were met according to RECIST 1.0 criteria.
Time Frame: as for outcome 2
Population: Patients from the Treated Set (TS) with objective response.
Measure: Median (Full Range); unit: days
Arm/Group | Afatinib 20mg With Vinorelbine i.v. | Afatinib 40mg With Vinorelbine i.v. | Afatinib 50mg With Vinorelbine i.v. | Afatinib 20mg With Vinorelbine Per os | Afatinib 40mg With Vinorelbine Per os | Afatinib 50mg With Vinorelbine Per os
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 3 | 0
days |  |  |  |  | 55 [55 to 343] |

6. Secondary Outcome: Duration of Objective Response
Description: The duration of objective response was measured from the time of first documented confirmed CR or PR to the time of progressive disease or death, whichever occured earlier.
Time Frame: as for outcome 2
Population: Patients from Treated Set (TS) with Objective Response.
Measure: Median (Full Range); unit: days
Arm/Group | Afatinib 20mg With Vinorelbine i.v. | Afatinib 40mg With Vinorelbine i.v. | Afatinib 50mg With Vinorelbine i.v. | Afatinib 20mg With Vinorelbine Per os | Afatinib 40mg With Vinorelbine Per os | Afatinib 50mg With Vinorelbine Per os
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 3 | 0
days |  |  |  |  | 114 [113 to 151] |

7. Secondary Outcome: Duration of Disease Control
Description: Duration of disease control was measured from the start of study treatment to the time of progression or death, whichever occured first.
Time Frame: as for outcome 2
Population: Patients from Treated Set (TS) with disease control.
Measure: Median (Full Range); unit: days
Arm/Group | Afatinib 20mg With Vinorelbine i.v. | Afatinib 40mg With Vinorelbine i.v. | Afatinib 50mg With Vinorelbine i.v. | Afatinib 20mg With Vinorelbine Per os | Afatinib 40mg With Vinorelbine Per os | Afatinib 50mg With Vinorelbine Per os
Number analyzed (Participants) | 1 | 10 | 5 | 0 | 9 | 5
days | 110 [110 to 110] | 167 [94 to 351] | 168 [81 to 202] |  | 162 [50 to 493] | 120 [54 to 230]

8. Secondary Outcome: Best Percentage Change in Tumour Size
Description: Best percentage change in tumour size was the best percentage change in the sum of diameters of target lesions and was calculated as (minimum sum of diameters post baseline - sum of diameters at baseline)/sum of diameters at baseline. Negative values indicate a decrease, positive values an increase.
Time Frame: Screening and every 8 weeks after starting of treatment, up to 44 weeks.
Population: Patients from Treated Set (TS).
Measure: Mean (Standard Error); unit: percentage change in tumour size
Arm/Group | Afatinib 20mg With Vinorelbine i.v. | Afatinib 40mg With Vinorelbine i.v. | Afatinib 50mg With Vinorelbine i.v. | Afatinib 20mg With Vinorelbine Per os | Afatinib 40mg With Vinorelbine Per os | Afatinib 50mg With Vinorelbine Per os
Number analyzed (Participants) | 3 | 19 | 6 | 4 | 18 | 5
percentage change in tumour size | -5.65 (10.91) | -7.51 (4.22) | -24.10 (9.57) | 25.89 (4.55) | -1.36 (9.62) | -10.76 (3.47)

9. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from the first dose of study medication to the occurrence of tumour progression or death, whichever came first. It was assessed according to RECIST 1.0. Median time results from unstratified Kaplan-Meier estimates.
Time Frame: From first dose of study medication to the occurrence of progression or death whichever came first, up to 44 months.
Population: All patients treated in the MTD cohorts.
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Afatinib 40mg With Vinorelbine i.v. | Afatinib 40mg With Vinorelbine Per os
Number analyzed (Participants) | 19 | 18
weeks | 14.6 [7.1 to 31.9] | 15.9 [7.4 to 23.7]

10. Secondary Outcome: Area Under the Concentration-time Curve of Afatinib After Multiple Administrations of 40mg Afatinib in Presence and Absence of 25mg/m^2 i.v. Vinorelbine at Steady State
Time Frame: 0.05 hours (h) before dosing at day 1 and 0.10h, 0.30h, 1h, 4h, 7h, 24h and 168h after dosing, 0.05 hours (h) before dosing at day 15 and day 21 and 0.10h, 0.30h, 1h, 2h, 3h, 4h, 6h, 7h and 24h after dosing
Population: All patients treated in the MTD cohort, for which evaluable PK parameters were available for the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- in Presence of Vinorelbine i.v.: Afatinib 40 mg in presence of 25mg/m^2 vinorelbine i.v.
- in Absence of Vinorelbine i.v.: Afatinib 40 mg in absence of 25mg/m^2 vinorelbine i.v.
Arm/Group | in Presence of Vinorelbine i.v. | in Absence of Vinorelbine i.v.
Number analyzed (Participants) | 14 | 8
ng*h/mL | 892 (87.3) | 683 (375.0)
Statistical Analysis 1: Comparison: in Presence of Vinorelbine i.v. vs in Absence of Vinorelbine i.v; Test type: Superiority or Other; ANOVA; Ratio of adjusted gMean = 126.20, 90% CI 2-sided [69.549 to 229.012]

11. Secondary Outcome: Area Under the Concentration-time Curve of Vinorelbine After Single and Multiple Intravenous Administrations of 25mg/m^2 Vinorelbine in Presence and Absence of Afatinib at Steady State
Time Frame: as for outcome 10
Population: All patients treated in the TS, for which evaluable PK parameters were available for the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- in Presence of Afatinib: 25mg/m^2 vinorelbine i.v. in presence of Afatinib 20, 40 and 50 mg
- in Absence of Afatinib: 25mg/m^2 vinorelbine i.v. in absence of Afatinib 20, 40 or 50 mg
Arm/Group | in Presence of Afatinib | in Absence of Afatinib
Number analyzed (Participants) | 12 | 18
ng*h/mL | 512 (41.4) | 655 (26.0)
Statistical Analysis 1: Comparison: in Presence of Afatinib vs in Absence of Afatinib; Test type: Superiority or Other; ANOVA; Ratio of adjusted gMean = 75.58, 90% CI 2-sided [65.037 to 87.837]

12. Secondary Outcome: Maximum Measured Concentration of Afatinib After Multiple Administrations of 40mg Afatinib in Presence and Absence of 25mg/m^2 i.v. Vinorelbine at Steady State
Time Frame: as for outcome 10
Population: All patients treated in the MTD cohort, for which evaluable PK parameters were available for the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | in Presence of Vinorelbine i.v. | in Absence of Vinorelbine i.v.
Number analyzed (Participants) | 14 | 8
ng/mL | 62.0 (97.9) | 42.7 (425)
Statistical Analysis 1: Comparison: in Presence of Vinorelbine i.v. vs in Absence of Vinorelbine i.v; Test type: Superiority or Other; ANOVA; Ratio of adjusted gMean = 132.80, 90% CI 2-sided [72.305 to 243.917]

13. Secondary Outcome: Maximum Measured Concentration of Vinorelbine After Single and Multiple Intravenous Administrations of 25 mg/m^2 Vinorelbine in Presence and Absence of Afatinib at Steady State
Time Frame: as for outcome 10
Population: All patients treated in the TS, for which evaluable PK parameters were available for the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- in Presence of Afatinib: 25mg/m^2 vinorelbine i.v. in presence of Afatinib 20, 40 and 50mg Afatinib
- in Absence of Afatinib: 25mg/m^2 vinorelbine i.v. in absence of Afatinib 20, 40 and 50mg Afatinib
Arm/Group | in Presence of Afatinib | in Absence of Afatinib
Number analyzed (Participants) | 12 | 18
ng/mL | 822 (56.2) | 941 (55.1)
Statistical Analysis 1: Comparison: in Presence of Afatinib vs in Absence of Afatinib; Test type: Superiority or Other; ANOVA; Ratio of adjusted gMean = 83.80, 90% CI 2-sided [61.156 to 114.823]

14. Secondary Outcome: Time From Dosing to the Maximum Concentration of Afatinib After Multiple Administrations of 40mg Afatinib in Presence and Absence of 25mg/m^2 i.v. Vinorelbine at Steady State
Time Frame: as for outcome 10
Population: All patients treated in the MTD cohort, for which evaluable PK parameters were available for the analysis.
Measure: Median (Full Range); unit: hours
Arm/Group | in Presence of Vinorelbine i.v. | in Absence of Vinorelbine i.v.
Number analyzed (Participants) | 14 | 8
hours | 3.16 [2.00 to 6.00] | 2.00 [1.00 to 4.03]

15. Secondary Outcome: Time From Dosing to the Maximum Concentration of Vinorelbine After Single and Multiple Intravenous Administrations of 25mg/m^2 Vinorelbine in Presence and Absence of Afatinib at Steady State
Time Frame: as for outcome 10
Population: All patients treated in the TS, for which evaluable PK parameters were available for the analysis.
Measure: Median (Full Range); unit: hours
Arm/Group | in Presence of Afatinib | in Absence of Afatinib
Number analyzed (Participants) | 12 | 18
hours | 0.166 [0.150 to 0.167] | 0.167 [0.150 to 0.233]

16. Secondary Outcome: Area Under the Concentration-time Curve of Afatinib After Multiple Administrations of 40mg Afatinib in Presence and Absence of 60mg/m^2 Per os Vinorelbine at Steady State
Time Frame: 0.05 hours (h) before dosing at day 1 and 1h, 1.30h, 2h, 3h, 6h,, 7h and 24h after dosing
Population: All patients treated in the MTD cohort, for which evaluable PK parameters were available for the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- in Presence of Vinorelbine Per os: Afatinib 40 mg in presence of 60mg/m^2 vinorelbine per os.
- in Absence of Vinorelbine Per os: Afatinib 40 mg in absence of 60mg/m^2 vinorelbine per os.
Arm/Group | in Presence of Vinorelbine Per os | in Absence of Vinorelbine Per os
Number analyzed (Participants) | 9 | 8
ng*h/mL | 872 (39.8) | 1070 (33.8)
Statistical Analysis 1: Comparison: in Presence of Vinorelbine Per os vs in Absence of Vinorelbine Per os; Test type: Superiority or Other; ANOVA; Ratio of adjusted gMean = 90.21, 90% CI 2-sided [76.071 to 106.978]

17. Secondary Outcome: Area Under the Concentration-time Curve of Vinorelbine After Multiple Administrations Per os of 60mg/m^2 Vinorelbine in Presence and Absence of Afatinib at Steady State
Time Frame: 0.05 hours (h) before dosing at day 1 and 1h, 1.30h, 2h, 3h, 6h, 7h and 24h after dosing
Population: All patients treated in the TS, for which evaluable PK parameters were available for the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- in Presence of Afatinib: 60 mg/m^2 vinorelbine per os in presence of Afatinib
- in Absence of Afatinib: 60 mg/m^2 vinorelbine per os in absence of Afatinib
Arm/Group | in Presence of Afatinib | in Absence of Afatinib
Number analyzed (Participants) | 15 | 25
ng*h/mL | 258 (79.8) | 334 (70.9)
Statistical Analysis 1: Comparison: in Presence of Afatinib vs in Absence of Afatinib; Test type: Superiority or Other; ANOVA; Ratio of adjusted gMean = 76.75, 90% CI 2-sided [56.710 to 103.871]

18. Secondary Outcome: Maximum Measured Concentration of Afatinib After Multiple Administrations of 40mg Afatinib in Presence and Absence of 25mg/m^2 Per os Vinorelbine at Steady State
Time Frame: 0.05 hours (h) before dosing at day 1 and 1h, 1.30h, 2h, 3h, 6h, 7h and 24h after dosing
Population: All patients treated in the MTD cohort, for which evaluable PK parameters were available for the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- in Presence of Vinorelbine Per os: Afatinib 40 mg in presence of 25mg/m^2 vinorelbine per os
- in Absence of Vinorelbine Per os: Afatinib 40 mg in absence of 25mg/m^2 vinorelbine per os
Arm/Group | in Presence of Vinorelbine Per os | in Absence of Vinorelbine Per os
Number analyzed (Participants) | 10 | 9
ng/mL | 55.1 (35.6) | 67.2 (29.4)
Statistical Analysis 1: Comparison: in Presence of Vinorelbine Per os vs in Absence of Vinorelbine Per os; Test type: Superiority or Other; ANOVA; Ratio of adjusted gMean = 83.86, 95% CI 2-sided [66.369 to 105.966]

19. Secondary Outcome: Maximum Measured Concentration of Vinorelbine After Multiple Administrations Per os of 60mg/m^2 in Presence and Absence of Afatinib at Steady State
Time Frame: as for outcome 10
Population: All patients treated in the TS, for which evaluable PK parameters were available for the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- in Presence of Afatinib: 60mg/m^2 vinorelbine per os in presence of afatinib
- in Absence of Afatinib: 60mg/m^2 vinorelbine per os in absence of afatinib
Arm/Group | in Presence of Afatinib | in Absence of Afatinib
Number analyzed (Participants) | 15 | 25
ng/mL | 52.8 (80.8) | 65.0 (63.9)
Statistical Analysis 1: Comparison: in Presence of Afatinib vs in Absence of Afatinib; Test type: Superiority or Other; ANOVA; Ratio of adjusted gMean = 81.70, 90% CI 2-sided [60.470 to 110.369]

20. Secondary Outcome: Time From Dosing to the Maximum Concentration of Afatinib After Multiple Administrations of 40mg Afatinib in Presence and Absence of 60mg/m^2 Per os Vinorelbine at Steady State
Time Frame: 0.05 hours (h) before dosing at day 1 and 1h, 1.30h, 2h, 3h, 6h, 7h and 24h after dosing
Population: All patients treated in the MTD cohort, for which evaluable PK parameters were available for the analysis.
Measure: Median (Full Range); unit: hours
Arm/Group | in Presence of Vinorelbine Per os | in Absence of Vinorelbine Per os
Number analyzed (Participants) | 10 | 9
hours | 3.54 [2.00 to 5.03] | 3.00 [1.00 to 6.00]

21. Secondary Outcome: Time From Dosing to the Maximum Concentration of Vinorelbine After Single and Multiple Administrations of 60mg/m^2 Vinorelbine Per os in Presence and Absence of Afatinib at Steady State
Time Frame: 0.05 hours (h) before dosing at day 1 and 1h, 1.30h, 2h, 3h, 6h, 7h and 24h after dosing
Population: All patients treated in the TS, for which evaluable PK parameters were available for the analysis.
Measure: Median (Full Range); unit: hours
Arm/Group | in Presence of Afatinib | in Absence of Afatinib
Number analyzed (Participants) | 15 | 25
hours | 1.50 [1.00 to 6.00] | 1.50 [0.917 to 3.17]

ADVERSE EVENTS:
Time Frame: First administration of trial medication until 28 days after last administration of trial medication.
Groups:
- Afatinib 20mg With Vinorelbine i.v.: Continuous daily dosing of Afatinib 20mg orally and weekly Vinorelbine 25 mg/m2 intravenously (days 1, 8, 15 and 22) in a 4-weekly course. Patients will be eligible for repeated treatment courses in the absence of clinical disease progression or undue toxicity .
- Afatinib 40mg With Vinorelbine i.v.: Continuous daily dosing of Afatinib 40mg orally and weekly Vinorelbine 25 mg/m2 intravenously (days 1, 8, 15 and 22) in a 4-weekly course. Patients will be eligible for repeated treatment courses in the absence of clinical disease progression or undue toxicity .
- Afatinib 50mg With Vinorelbine i.v.: Continuous daily dosing of Afatinib 50mg orally and weekly Vinorelbine 25 mg/m2 intravenously (days 1, 8, 15 and 22) in a 4-weekly course. Patients will be eligible for repeated treatment courses in the absence of clinical disease progression or undue toxicity .
- Afatinib 40mg With Vinorelbine Per os: Continuous daily dosing of Afatinib 40mg orally and oral vinorelbine 60 mg/m2/week for days 1,8,15 of first cycle, and 80mg/m2 from day 22 first cycle onwards, weekly. Patients will be eligible for repeated treatment courses in the absence of clinical disease progression or undue toxicity .
- Afatinib 50mg With Vinorelbine Per os: Continuous daily dosing of Afatinib 50mg orally and oral vinorelbine 60 mg/m2/week for days 1,8,15 of first cycle, and 80mg/m2 from day 22 first cycle onwards, weekly. Patients will be eligible for repeated treatment courses in the absence of clinical disease progression or undue toxicity .
Arm/Group | Afatinib 20mg With Vinorelbine i.v. | Afatinib 40mg With Vinorelbine i.v. | Afatinib 50mg With Vinorelbine i.v. | Afatinib 20mg With Vinorelbine Per os | Afatinib 40mg With Vinorelbine Per os | Afatinib 50mg With Vinorelbine Per os
Serious Adverse Events (participants affected / at risk) | 1/3 | 11/19 | 4/6 | 2/4 | 13/18 | 1/5
Other Adverse Events (participants affected / at risk) | 3/3 | 19/19 | 6/6 | 4/4 | 18/18 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib 20mg With Vinorelbine i.v. (N=3) | Afatinib 40mg With Vinorelbine i.v. (N=19) | Afatinib 50mg With Vinorelbine i.v. (N=6) | Afatinib 20mg With Vinorelbine Per os (N=4) | Afatinib 40mg With Vinorelbine Per os (N=18) | Afatinib 50mg With Vinorelbine Per os (N=5)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 3 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 2 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 1 | 0 | 2 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 2 | 1
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
General physical health deterioration (General disorders) | 1 | 0 | 0 | 0 | 2 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 1 | 0 | 1 | 0
Hepatocellular injury (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Biliary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Aphasia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hemianopia homonymous (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Intracranial pressure increased (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib 20mg With Vinorelbine i.v. (N=3) | Afatinib 40mg With Vinorelbine i.v. (N=19) | Afatinib 50mg With Vinorelbine i.v. (N=6) | Afatinib 20mg With Vinorelbine Per os (N=4) | Afatinib 40mg With Vinorelbine Per os (N=18) | Afatinib 50mg With Vinorelbine Per os (N=5)
Anaemia (Blood and lymphatic system disorders) | 1 | 9 | 3 | 2 | 8 | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 1 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 3 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 12 | 3 | 1 | 8 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Atrioventricular block (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Ear disorder (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 1 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 1 | 0 | 1 | 0
Blepharitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 1
Dry eye (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 0
Exophthalmos (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Eyelid ptosis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Lacrimation increased (Eye disorders) | 0 | 1 | 0 | 1 | 1 | 0
Ocular icterus (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Photopsia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 3 | 2 | 1 | 5 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 5 | 1 | 1 | 2 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Anorectal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 4 | 1 | 0 | 1 | 2
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Chapped lips (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 1 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 7 | 2 | 2 | 7 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 19 | 6 | 2 | 17 | 5
Dry mouth (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 1 | 1 | 1 | 3 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 4 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 4 | 1
Gingival bleeding (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 1 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 3 | 1 | 1 | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 12 | 5 | 3 | 11 | 4
Odynophagia (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Portal hypertensive gastropathy (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 7 | 2 | 0 | 7 | 2
Tongue ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 8 | 4 | 1 | 13 | 3
Asthenia (General disorders) | 2 | 19 | 6 | 4 | 14 | 5
Catheter site pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 2 | 0 | 0 | 2 | 2
Chills (General disorders) | 1 | 0 | 0 | 1 | 0 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Feeling cold (General disorders) | 0 | 2 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Hyperthermia (General disorders) | 0 | 0 | 0 | 0 | 2 | 0
Inflammation (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Mucosal discolouration (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 8 | 4 | 0 | 6 | 2
Oedema peripheral (General disorders) | 1 | 3 | 2 | 0 | 2 | 1
Pain (General disorders) | 0 | 2 | 0 | 0 | 0 | 1
Puncture site pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 10 | 2 | 2 | 6 | 2
Ulcer (General disorders) | 0 | 2 | 0 | 0 | 2 | 0
Xerosis (General disorders) | 0 | 2 | 1 | 1 | 1 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 3 | 0 | 1 | 2 | 0
Hepatocellular injury (Hepatobiliary disorders) | 0 | 6 | 1 | 0 | 2 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Escherichia infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Folliculitis (Infections and infestations) | 0 | 7 | 2 | 0 | 7 | 2
Fungal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Fungal oesophagitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Fungal paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Furuncle (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Genital infection fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Herpes virus infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Lymphangitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 3 | 2 | 0 | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Oral fungal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 2
Otitis externa (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 5 | 2 | 0 | 5 | 3
Pharyngitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0
Proteus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pulpitis dental (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Puncture site abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0
Rhinitis (Infections and infestations) | 0 | 6 | 3 | 0 | 4 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 2 | 0 | 0 | 1 | 0
Tinea pedis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0
Upper respiratory fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 4 | 0 | 0 | 1 | 1
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection enterococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Burn oesophageal (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Amylase increased (Investigations) | 0 | 2 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0 | 2 | 1
Blood phosphorus decreased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0
Eastern Cooperative Oncology Group performance status worsened (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 4 | 3 | 2 | 2 | 2
White blood cell count increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 1
Cell death (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 13 | 4 | 3 | 10 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 3 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hyperproteinaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 2 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 5 | 3 | 0 | 5 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0 | 0 | 4 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 5 | 3 | 0 | 4 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1 | 0 | 3 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 1 | 1 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Sarcopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Haemangioma of bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Aphonia (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cerebral microhaemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cervical root pain (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dysaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 4 | 2 | 0 | 2 | 2
Epilepsy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 2 | 1 | 0 | 2 | 1
Hydrocephalus (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 2 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 4 | 5 | 1 | 5 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Sensory loss (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 2 | 1 | 1 | 0 | 0
Toxic neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 2 | 2 | 4 | 3
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 2 | 1
Hallucination, visual (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 2 | 2 | 1
Sleep disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Bladder discomfort (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 2 | 1 | 0 | 1 | 1
Micturition disorder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Genital lesion (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Genital tract inflammation (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Scrotal oedema (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 9 | 2 | 1 | 4 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 1 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 9 | 2 | 0 | 7 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 4 | 0 | 4 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0 | 0 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 4 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 4 | 2 | 0 | 2 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 4 | 1 | 1 | 4 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 4 | 1 | 0 | 1 | 0
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nail pigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nail pitting (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0
Nail toxicity (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 7 | 1 | 0 | 9 | 3
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 3 | 2 | 0 | 3 | 3
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Xeroderma (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 2 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 1 | 0 | 1 | 0
Intermittent claudication (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Lymphoedema (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pallor (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.